CLINICAL TRIAL: NCT04378894
Title: Randomized Controlled Trial and Process Evaluation of the Mother-Child Educational Program (MOCEP) in Riyadh, Saudi Arabia.
Brief Title: Evaluation of the Mother-Child Educational Program (MOCEP) in Riyadh, Saudi Arabia.
Acronym: MOCEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Maha Muneef, professor of pediatrics infectious Diseases, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC17/259/R
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Parenting
Keywords: MOCEP, Parenting, Saudi Arabia

STUDY DESIGN:
Intervention Model Description: Randomized wait-list controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The mothers in the control group will take a special awareness program but not MOCEP and the participant, the care providers and the investigators are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOCEP (Experimental): MOCEP is implemented over a period of 25 weeks, through weekly group meetings that last approximately three hours.
  Interventions: Behavioral: MOCEP
- Waitlist Control Group (Active Comparator): For ethical reasons, no one recruited will be excluded from the opportunity to benefit from the intervention. MOCEP group will be the primary intervention group and the second group will act as the wait-listed control group. Families in the wait-listed control group will participate in a special awareness program but not MOCEP. Although the families in the wait-listed control group will start as a control group (not receiving the intervention), they will have the opportunity to participate in the intervention in a later round of implementation, after the intervention group has completed the program.
  Interventions: Behavioral: MOCEP

INTERVENTIONS:
Behavioral: MOCEP — Through parent support and an evidence-based curriculum, MOCEP uses education to reduce risk factors that hinder children's health and wellbeing.

SUMMARY:
The Mother Child Education Program (MOCEP) was developed by the Mother Child Education Foundation (ACEV). MOCEP is implemented in Saudi Arabia through a 25-week program conducted by ACEV-trained groups with a curriculum for the child that is implemented at home by the mothers. The program is designed to (1) promote parenting skills and bolster strategies that support school readiness among mothers of 3-to-6- year-old children, and (2) enhance social cohesion in the family and community. Rigorous evaluations of MOCEP have been conducted in several contexts, but not yet in the context of Saudi Arabia. Thus, the present study aims to rigorously evaluate the impact of MOCEP on child and parent outcomes among families in Riyadh, Saudi Arabia.

DETAILED DESCRIPTION:
The problem and its importance: According to an estimate two hundred million or a third of the world's youngest children do not achieve their potential due to lack of stimulating, nurturing, safe, and responsive caregiving. The importance of caregiving cannot be underestimated for early child development (Engle et al.,2007). However, parents and caregivers need to be supported in fulfilling this role. The results from parenting programs, across high-, middle and low-income countries indicate significant trends in obtaining positive results for parents and children (MOCEP).

In Saudi Arabia, youth represents almost 50% of the population and those < 5 years of age account for 10.6% (GaStat, 2019). As for the crude birth rate among the Saudi population, it hits 17.23 live children for every 1,000 persons. Thus, the government has stressed the importance of investing in national programs that focus on childhood within the scope of the 2030 vision. MOCEP was implemented in Saudi Arabia by the Child Care Association (CCA) which is an NGO established in 2006. The CCA's main objective is to promote Early Child Development (ECD) through the MOCEP since 2011.

The purpose of the present evaluation study--a collaboration between CCA and KAIMRC--is to evaluate the impact of MOCEP on child and parent outcomes among families in Riyadh, Saudi Arabia, using a randomized wait-list controlled trial. Specifically, the aim of the study is to empirically assess the impact of MOCEP on maternal and child outcomes and to explore key moderators of the programmatic impact including characteristics of the program implementation and contextual characteristics.

Specific Objective 1: We will characterize the impact of MOCEP on child outcomes including executive function, social-emotional skills, and cognitive skills such as emergent numeracy, literacy and verbal skills.

Specific Objective 2: We will characterize the impact of MOCEP on parental knowledge, attitudes, practices, and skills.

A comprehensive sociodemographic characterization of participating mothers and children will be conducted. Maternal and child outcomes will be measured before and after the intervention. Maternal outcomes will include knowledge, attitudes, and practices regarding parenting, child development, and education; disciplinary style; wellbeing; social support; and empowerment. Child outcomes will include executive function, social-emotional skills, nutritional status, and school readiness. Mothers will complete a demographic questionnaire at baseline to characterize social, demographic, home, family, and community characteristics. Mothers will also complete a battery addressing parenting and child development-related knowledge, attitudes and practices at baseline and endline.

The assessors will use IDELA which provides a direct measure of children's learning and development and assesses child school readiness through a holistic exploration of children's early literacy, math, problem-solving, social-emotional development, and gross and fine motor skills. The tool is available in Arabic and has been validated in multiple countries.

To assess the social-emotional skills of children, in addition to the IDELA subtest, we will apply the Strengths and Difficulties Questionnaire. This parent-report measure assesses children's emotional and conduct problems, hyperactivity, and peer relations.

The Disciplinary Style Questionnaire (DSQ), a parent-report measure of parental disciplinary style, will be used to assess the frequency with which parents engage in seven forms of discipline when dealing with children's undesirable behavior: inductive discipline, physical punishment, manipulating privileges, harsh verbal discipline, argument, shaming, and ignoring. These outcomes will be measured before and after implementation of the 25 weeks MOCEP program.

Process evaluation:

Program dosage: will be measured by mothers' attendance at training sessions and the number of sessions delivered by group leaders will be collected using attendance sheets.

Program engagement: will be measured by a set of items that will be developed by the Yale study team, based on constructs examined in other studies (Durlak & DuPre, 2008; Reyes et aL, 2012). The tool measuring program engagement will be administered to both parents and group leaders participating in MOCEP.

Program quality: will be measured with observational tools and self-report measures. An ethnographer will be present during the training to document facets such as trainer responsiveness to parents' needs, clarity of delivery, trainer motivation, parent engagement, and group cohesion. Also, supervisors will complete the MOCEP Supervisor's Checklist; supervisors and parents will rate the overall quality of training using items developed by the research team. Finally, MOCEP curriculum worksheets will be used to determine the degree to which mothers deliver the program as intended in their homes.

Data will be collected in paper forms by trained assessors and then entered into a secured electronic database prepared by KAIMRC using the KoBo Toolbox program.

Sample size: We aim to recruit 100 mother-child dyads for the wait-list control and 100 mother-child dyads for the intervention group.

Sampling technique: The target population will be recruited based on the catchment areas for the program in the Riyadh area (convenience sampling). We will randomize the enrolled participants to the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Mothers must have at least one child between 3 and 6 years of age.
* Mothers must be literate.
* Mothers must be living in the designated implementation areas in Riyadh, Saudi Arabia.
* Mothers must agree to attend the MOCEP program and complete questionnaires at the beginning and the end of the program

Exclusion Criteria:

• No signed consent

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Disciplinary Style Questionnaire | 25 weeks
  Parent report measure of parental disciplinary style assesses the frequency with which parents engage in seven forms of discipline when dealing with children's undesirable behavior
Better Parenting Questionnaire | 25 weeks
  11-item questionnaire that measures responsive parenting as reported by the mother
International Development and Early Learning Assessment (IDELA) | 25 weeks
  An, easy-to-use, rigorous global tool that measures children's early learning and development of children from 3.5 to 6 years of age.

SECONDARY OUTCOMES:
Social-Emotional Status: Strengths and Difficulties Questionnaire (child assessment) | 25 weeks
  Parent report measure assesses children's emotional and conduct problems, hyperactivity, and peer relations.
Parenting Stress Index (PSI) | 25 weeks
  36-item questionnaire that measures maternal perceptions of stress in the role of a parent.
Individual Distress Assessment (IDA) | 25 weeks
  Mothers are asked to report the extent to which they are currently feeling a number of affects (e.g., frustrated, lonely, anxious) using this 12-item rating scale.
Father Involvement Questionnaire (FIQ) | 25 weeks
  20 items that measure the mothers' perceptions of how her husband interacts with their children, how the mother is treated by her husband, and how her husband interacts with other members of the community.

CONTACTS AND LOCATIONS:
Overall Officials: majid aljeraisy, PHD, Study Chair — riyadh , saudi arabia
Locations (1):
- Woman and Child Association, Riyadh, Saudi Arabia